CLINICAL TRIAL: NCT06161272
Title: A Randomized, Multicenter, Noncomparative Clinical Study of Fluzoparib With or Without Apatinib for Maintenance Therapy in PARPi-pretreated Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: Fluzoparib With or Without Apatinib in Platinum-sensitive Relapsed Ovarian Cancer Previously Treated With PARPi
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Li Li, Prof., Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS2023(166)
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; High Grade Serous Adenocarcinoma of Ovary; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
Keywords: ovarian cancer; PARP inhibitors; Flzuoparib; Antiangiogenic agents; Apatinib
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1：Fluzoparib (Experimental): Fluzoparib capsule: oral administration, 3 capsules/dose (150 mg/ dose), twice a day, in the morning and evening, before/after meals can be taken orally, it is recommended to take orally within 0.5h after breakfast and dinner, continuous administration. Every 4 weeks is a treatment cycle.
  Interventions: Drug: Fluzoparib
- Arm2：Fluzoparib + apatinib (Experimental): Fluzoparib capsule: oral administration, 2 capsules/dose (100 mg/ dose), twice a day, in the morning and evening, before/after meals can be taken orally, it is recommended to take orally within 0.5h after breakfast and dinner, continuous administration. Every 4 weeks is a treatment cycle.
  Apatinib: oral administration, 1 tablet/dose (375 mg/tablet), once a day, it is recommended to take orally within 0.5h after breakfast, continuous administration. Every 4 weeks is a treatment cycle.
  Interventions: Drug: Fluzoparib+Apatinib

INTERVENTIONS:
Drug: Fluzoparib — single
  Arms: Arm1：Fluzoparib
Drug: Fluzoparib+Apatinib — combination
  Arms: Arm2：Fluzoparib + apatinib

SUMMARY:
This is a randomized, multicenter, two-arm, noncomparative, phase II study of fluzoparib with or without apatinib for maintenance therapy in PARPi-pretreated platinum-sensitive recurrent ovarian cancer. The primary objective is to evaluate median progression free survival of fluzoparib with or without apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined the study and signed the informed consent.
2. Female, 18-75 years (calculated on date of signing informed consent).
3. Participant has histologically confirmed diagnosis of high-grade predominantly serous ovarian cancer, fallopian tube cancer, primary peritoneal cancer; ≥grade II ovarian endometrioid adenocarcinoma.

   - Mixed tumors: contain high-grade serous component or endometrioid components over 50%.
4. Disease progression greater than 6 months (184 days) after completion of their last dose of platinum chemotherapy.
5. Prior treatment with ≥2 platinum-containing chemotherapy regimens and disease remission (complete or partial response) at the end of the last platinum chemotherapy, which lasted until study administration, must be randomized to enrollment and start trial drug administration within 8 weeks from the last chemotherapy administration.

   * Preoperative neoadjuvant chemotherapy and postoperative chemotherapy counted as 1 chemotherapy treatment regimen.
   * The last chemotherapy must be a platinum-based chemotherapy regimen.
   * Patient must have received at least 4 cycles of treatment for the last platinum-based chemotherapy, during or after platinum-containing chemotherapy, concurrent use of other investigational drugs and treatment other than endocrine therapy drugs are not permitted.
   * A detectable lesion or CA-125 ≥2 ×ULN is required before the last platinum treatment.
   * The imaging results showed CR or PR during the last platinum-containing regimen, CA125 decreased to within the ULN or ≥90% from pre-treatment level during treatment and CA125 remained <1xULN or did not increase by >10% in 7 days before the first treatment.
   * If no lesion is assessed prior to chemotherapy, CA125 should be alleviated to the ULN during treatment and maintained at <1xULN for 7 days prior to the first treatment.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. The duration of continuous PARPi treatment during the previous maintenance treatment period was ≥6 months.
8. Participant has adequate organ function as defined in the following contents (Any blood component or cell growth factor within 14 days prior to randomization is not permitted)

   * Absolute neutrophil count (ANC) ≥1.5×10^9/L
   * Platelets ≥100×10^9/L
   * Hemoglobin ≥9g/dL
   * Serum albumin ≥3g/dL
   * Total bilirubin ≤1.5 ×ULN
   * AST and ALT ≤3 × ULN, and for patients with liver metastases, AST and ALT levels ≤5× ULN
   * Serum creatinine ≤1.5 × ULN.
9. Patients with potential fertility must have had a negative blood or urine pregnancy test within 72 hours prior to the first dose, are not breastfeeding, and must agree to use a medically approved contraceptive (e.g., intrauterine device, birth control pill or condom) for the duration of the trial and for a period of 6 months after the last administration of fluzoparib or 2 months after the last administration of apatinib, whichever is longer.

Exclusion Criteria:

1. Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry; Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix or breast cancer without recurrence over 3 years allowed.
2. The expected survival is less than three months.
3. Participants with untreated central nervous system metastases

   - patients who had previously received systemic, radical brain or meninges metastases (radiotherapy or surgery), had been stable for at least 1 month on imaging, had stopped systemic sex hormone therapy (dose >10mg/ day or other therapeutic hormones) for more than 2 weeks, and had no clinical evidence could be included.
4. Not able to swallow pills normally, or have abnormal gastrointestinal function affecting drug absorption as judged by the researcher.
5. Intestinal obstruction within 3 months.
6. The urine protein ≥ ++ and 24-hour urine protein level > 1.0g.
7. Patients with clinical symptoms of cancer ascites, pleural effusion, who need to drainage, or who have undergone ascites drainage within 2 months prior to the first administration.
8. Uncontrolled heart clinical symptoms or diseases, such as :(1) NYHA 2 or more heart failure, (2) Unstable angina pectoris, (3) myocardial infarction within 1 year, (4) Ventricular arrhythmias requiring intervention, (5) QTc>470ms.
9. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds), bleeding tendency or receiving thrombolytic therapy are allowed to receive low-dose low-molecular weight heparin or oral aspirin preventive anticoagulant therapy during the study.
10. Significant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis, etc., within the first 3 months of the randomization. If fecal occultation blood is positive at baseline, gastroscopy should be performed if still positive after reexamination.
11. Active ulcers, unhealed wounds or fractures.
12. Uncontrolled hypertension by antihypertensive medication (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥90mmHg).
13. Any bleeding event with grade 2 or higher in CTCAE 5.0 within 4 weeks prior randomization.
14. Active infection or unexplained fever >38.5 degrees during screening or before first treatment.
15. Participants with congenital or acquired immune deficiency (such as HIV infection), or active hepatitis (hepatitis B reference: HBsAg positive, HBV DNA≥500 IU/ml; Hepatitis C reference: HCV antibody positive, HCV virus copy number > upper limit of normal).
16. Received radiotherapy, chemotherapy, hormone therapy, or molecular targeted therapy, less than 4 weeks after the completion of the last dose or less than 5 drug half-lives before the study for oral molecular targeted drug; adverse events caused by previous treatment (except hair loss) and not recover to ≤1 degree (CTCAE 5.0).
17. Arteriovenous thrombosis events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. occurred within 6 months.
18. History of hereditary or acquired bleeding or coagulation disorders (e.g., hemophilia, coagulopathy, thrombocytopenia, etc.).
19. Need receive other systemic anti-tumor therapy during the study period.
20. According to the investigators' judgment the subjects had other factors that might have led to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | from the randomization up to 2 years
  Time from the date of randomization to the date of first documented tumor progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | from the randomization up to 3 years
  Time from the date of randomization to the date of death due to any cause.
Objective Response Rate (ORR) | from the randomization up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Disease control rate (DCR) | from the randomization up to two years
  the proportion of patients with a best overall response of confirmed complete or partial response or stable disease based on RECIST v1.1.
Time to start of first subsequent therapy or death (TFST) | from the randomization up to 3 years
  TFST is defined as the time from the randomization to the earliest of the date of anti-cancer therapy start date following study treatment discontinuation, or death.
Time to start of second subsequent therapy or death (TSST) | from the randomization up to 3 years
  TSST is defined as the time from the randomization to the earliest of the date of second subsequent anti-cancer therapy start date following study treatment discontinuation, or death.
Time to failure (TTF）by RECIST | from the randomization up to 3 years
  Time to treatment failure by RECIST v. 1.1 or CA-125 or death is defined as the time from the randomization to the date of RECIST progression or death by any cause, whichever occurs first.
Safety and tolerability | from the randomization up to 3 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Tumor Hospital of Guangxi Medical University., Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided